# Title:

Owning Rights and Protection: GBV Prevention, Mitigation, and Response in Colombia (2023-2025)

Date: February 27, 2024

NCT: NCT06312592

### **Contact email address**

a.harker@uniandes.edu.co

## **Project title**

Owning Rights and Protection: GBV Prevention, Mitigation, and Response in Colombia

# Investigador Principal (Profesor de la Universidad de los Andes)

Arturo Harker, PhD. Associate Professor at the School of Government, Universidad de Los Andes

## **Co-Principal Investigators**

Tatiana Andia, PhD. Professor at the Faculty of Social Sciences, Universidad de Los Andes

# **Students (specify project type: thesis, student initiative, other)**

None

# **Academic Unit of Principal Investigator**

Escuela de Gobierno, Universidad de los Andes

## Position of the principal investigator

Associate Professor

# **Financing entity**

- External
- □ Internal
- □ None other than my academic research workload

## Funding entity (specify institution, call, relevant academic unit)

United States' Bureau of Population, Refugees and Migration

#### **Abstract**

As of August 2021, Colombia hosts the vast majority of Venezuelan refugees and migrants (UNHCR, 2022). For vulnerabile refugees and migrants in Colombia, and especially for women, gender-based violence (GBV) is present during transit and continues in their new homes where xenophobia, lack of accessible and adequate services, lack of safe economic opportunities, and lack of information on access to services, further increase risk. Lack of livelihood opportunities also affect vulnerable refugees and migrants, especially women, with barriers to employment including lack of information; precarious working conditions with lower payments and longer working days with increasing risks of labor exploitation; xenophobia and discrimination; limited access to formal labor markets; lack of access to financial services, among others. To address these issues, we are conducting a randomized-controlled trial )RCT) of HIAS' Entrepreneurship School with Gender Lens (ESGL), a methodology that targets GBV survivors and women at-risk to help them develop business ideas, access needed support for the prevention of and response to GBV, exploitation and trafficking, and improve participants' overall self-reliance. The RCT will be conducted within four cities in Colombia; approximately 80 eligible participants will be enrolled in each city and randomized to a treatment or control arm in a 2:1 ratio. Survey questionnaires will be administered to participants at baseline, eight months following baseline (endline), and 3-4 months after endline. Outcomes of interest include household self-reliance, mental health, empowerment, decision-making, and GBV risk and knowledge.

### **Background and Rationale**

Colombia is a major host of forcibly displaced Venezuelans, currently with approximately 2.5 million vulnerabile refugees and migrants. Colombia also has over 6.7 million internally displaced persons (IDPs) due to historical conflicts and violence. For vulnerabile refugees and migrants in Colombia, GBV is present during transit and continues in their new homes where xenophobia, lack of accessible and adequate services, lack of safe economic opportunities, and lack of information on access to services, further increase risk.

HIAS/UNHCR's 2022 study found limited availability of shelters and lack of protection services in border areas, placing women at a higher risk of violence by organised crime and drug traffickers. An increase in registered cases of GBV has also been identified as well as a trend in sexual relationships between adult men and VRAM girls and young women, promising economic

stability, or access to regularisation to control their partners, exposing girls and young women to cycles of violence and other negative consequences such as early pregnancy.

Vulnerable refugees and migrants also face psychosocial effects from their migratory experience, such as depression and anxiety and are further impacted by scarce protective resources when arriving in Colombia. This negative impact is more pronounced for GBV survivors due to psychological effects of enduring GBV, including low self-esteem, depression, fear, anguish, guilt, and post-traumatic stress.

Along with existing limitations in local institutional capacity to respond in the protection, health and justice sectors, xenophobia and institutional violence challenge access to services for GBV survivors. At the same time, local authorities lack knowledge on GBV survivors' rights and the required procedures to guarantee appropriate services, indicating the need to strengthen local capacity.

Lack of livelihood opportunities also affect vulnerable refugees and migrants, especially women. HIAS' latest Labor Market and Capacity Assessment identifies numerous barriers to seeking employment, including barriers in terms of regularisation; lack of information; precarious working conditions with lower payments and longer working days with increasing risks of labor exploitation; xenophobia and discrimination; limited access to formal labor markets; lack of access to financial services, among others.

#### Intervention

HIAS will promote the incubation of businesses through its Entrepreneurship School with Gender Lens (ESGL), a methodology that targets GBV survivors and women at-risk to help them develop business ideas, access needed support for the prevention of and response to GBV, exploitation and trafficking, and improve participants' overall self-reliance. Participants will go through a general business curriculum, work on business plans and learn gender issues and ways to mitigate GBV risks. Upon training completion, participants are eligible to pitch their business idea to a panel of experts and receive \$800 of seed capital. They will also receive follow-up business advisory support for at least six months, focusing on access to markets and finance and building support networks, in order to continue building self-reliance.

The ESGL will include a mental health and psychosocial support module, contributing to participant self-sufficiency, resilience, and empowerment through skills development such as coping skills, problem-solving capabilities, self-esteem, self-efficacy, communication abilities, self-regulation, and leadership, aimed at strengthening their ability to generate dignified livelihoods.

### Study objective

This study will conduct a pilot-randomised controlled trial to evaluate the entrepreneurship curriculum. The evaluation has three primary objectives:

- 1. Evaluate the preliminary effectiveness of the entrepreneurship programming to improve household self-reliance, mental health, and empowerment for households where women members run businesses.
- 2. Examine the relationship between GBV risk and self-reliance among women refugees in the Colombian migration context.
- 3. Assess the feasibility and acceptability of the refugee self-reliance index as a measurement tool in programs that strengthen self-reliance pathways for women individuals.

## Methodology

### Overview

This pilot RCT will be conducted in Cali, Ipiales, Pasto, and Popayan, and will include a control group. Eligible participants will be randomized to the treatment or control arm and the study team will collect data from both the intervention and comparison groups at: 1) the program baseline, 2) the program endline (8 months post-baseline), and 3) follow-up 3-4 months after program completion.

## **Screening for Eligibility: Inclusion Criteria**

Using their database and a pre-screening tool, HIAS will identify potential participants who meet the following criteria: women, at least 18 years of age, at risk of GBV or ever experienced GBV, have a migratory permit (for migrants and refugees), are Colombian or Venezuelan, have been residing in Colombia for at least six months, and have an entrepreneur profile registered with HIAS. Individuals with the targeted characteristics will then be further screened for study eligibility using the Self-Reliance Index (SRI). First launched in 2020, the Self-Reliance Index (SRI) is the first-ever global tool for measuring the progress of refugee households toward self-reliance (Seff, Leeson, and Stark, 2021). Eligible participants must receive a score between 2 and 3.5 on the tool to be included in the study. This range of scores aims to capture women who are vulnerable, but who are in a stable enough situation to develop an income generating activity (meaning that they are not unhoused or in need of urgent humanitarian assistance), while still in need of financial support, training and GBV assistance. If a participant's score on the SRI falls outside of the specified range, they will be ineligible for further inclusion, thanked for their time, and removed from the study. Participants whose score falls within the specified range will be included in the study and further baseline data will be collected including information on mental health, empowerment, and safety.

## Subject Recruitment, enrolment and sample size

HIAS will use their database and the pre-screening tool to identify potentially eligible participants for the study. They will aim to identify approximately 90-100 potentially eligible women through

the pre-screening tool. Official enrollment, consenting, and formal assessment of eligibility will be carried out by the research team. Data collectors will obtain written consent from previously pre-screened women prior to administering the SRI. After administering the SRI, data collectors will immediately administer the remaining survey questionnaire modules for participants whose SRI scores fall within the eligible range of 2 to 3.5. Women whose scores fall outside of the 2-3.5 range will be thanked for their time and not assigned to an evaluation arm.

Participants will be recruited from four cities: Cali, Ipiales, Pasto, and Popayan. The study will aim to enrol 80 women in the study within each city, where participants will be randomly assigned to the intervention or control arm at a 2:1 ratio.. As such, 90-100 women will be identified as potential participants through the pre-screening tool to account for ineligibility during the SRI administration phase.

At the time of enrolment, participants will receive a unique study ID. Following enrolment and baseline data collection, participants will be randomly assigned to the control or treatment arm using a random number generator in Stata (a data analysis software). The unique study ID will be used to track participants over time for future points of data collection.

#### Consent

Prior to data collection, the researcher will explain the study purpose, procedures, potential risks, and safeguards, such as participant confidentiality and referrals for services, where necessary. The researcher will explain that participants may be assigned to take part in the intervention based on randomization but that non-selection for the intervention will not prevent them from later participation in HIAS programs. They will be informed that they may also be provided with a referral for other programs. The researcher will emphasize that participation is completely voluntary and that participants will not be penalized in any way for choosing not to participate. Researchers will also explain and emphasize that participating or not participating in the study is purely voluntary and will have no impact on their access to future HIAS programming. Prospective participants will also be told that they are free to withdraw from the study at any time and to refuse to answer some or all of the questions. Participants will be informed that their data may be used by the research team in the future. The researcher will encourage the interviewee to ask any questions about the study processes before consenting to participate in the study.

Participants may feel compelled to consent to the study in spite of the above-mentioned informed consent procedures. Potential power differentials between the participants and data collectors may result in inadvertent coercion to participate in the study. The research team will carefully analyze the context-specific factors that may result in participant coercion and discuss strategies for ensuring genuine informed consent. Some of the measures that may be used include:

• Build on existing staff experience with informed consent procedures in other projects.

- Intensive staff training on the importance of informed consent and procedures to minimize potential coercion. Such procedures may include careful explanation and repetition of the nature of voluntary consent (e.g., participation in the study will not affect access to services; participants are free to refuse to answer any questions or to withdraw from the study at any time). Participants will also be given time to consider their decision.
- Multiple opportunities for participants to ask questions throughout the informed consent process and subsequent data collection. Researchers will be trained to respond to frequently asked questions or concerns that participants may raise. Close collaboration with HIAS staff to avoid recruiting participants who may be unable to provide assent voluntarily due to mental health or cognitive disability.

#### **Data Collection**

Participant data will be collected at three time points: baseline (when participants are first enrolled in the study), eight months post-baseline (upon program completion), and three months following endline data collection (eleven months after baseline). Data collectors will be hired and trained by Los Andes and the RSRI team members using a combination of online learning modules and in-person training, which will cover the study tools, evaluation protocol, humanitarian principles and its current practice, safeguarding policies, Psychological First Aid (PFA) gender and GBV, and research ethics and best practice.

## **Study Outcome Measures and Ascertainment**

#### Self-reliance:

The Self-Reliance Index (SRI) is the first-ever global tool for measuring the progress of refugee households toward self-reliance (Seff, Leeson, and Stark, 2021). The tool contains twelve domains focused on a household's basic needs, resources, and sustainability. Domains measure conditions and assets that increase the likelihood that refugees will be able to continue meeting their needs in the future. The study participant will respond on behalf of her household. The final self-reliance score may take a value from 1 to 5, with higher scores reflecting greater self-reliance. The tool is available in Spanish and has been previously validated with Venezuelan migrants in Colombia.

#### Resilience:

The Brief Resilient Coping Scale (BRCS) captures tendencies to cope adaptively with stress. The scale focuses on the tendency to effectively use coping strategies in a flexible and committed manner to actively solve problems despite stressful circumstances (Trejos Herrera et al., 2023).

Women's empowerment

Women's empowerment will be measured using the Women's Multidimensional Empowerment Index, which was developed using the 2015 Colombian Demographic and Health Survey (Rodríguez Guerrero, Nimeh, & Franco Correa, 2021). The index assesses empowerment multidimensionally based on the definition of empowerment proposed by Kabeer (1999) (Resources, domestic decision making, decision making on personal matters, and achievements), while capturing the notion of disempowerment.

Gender-based violence: Three items from the HIAS Knowledge and Perception of GBV risks and Women's Empowerment tool will be used. The HIAS tool was adapted based on other tools used in the Latin American region (cite). The three items pertain to self-reported perceptions of feeling supported by the community, feeling useful, and feeling controlled by one or more people. Responses are on a likert scale.

## **Ethical considerations**

### **Risks and Benefits**

According to Resolution number 008430 of 1993 of the Colombian Ministry of Health and Social Protection, this is "research without risk", which includes: "studies that employ retrospective documentary research techniques and methods and those in which no intervention or intentional modification of the biological, physiological, psychological or social variables of the individuals participating in the study is carried out, including: review of medical records, interviews, questionnaires and others in which no sensitive aspects of their behaviour are identified or dealt with".

The study is expected to carry minimal risk of loss of confidentiality associated with participation in group discussions, which will be minimized by data confidentiality measures and by using verbal informed consent procedures. Individuals have the option to not participate, or if they choose to participate, to decline to answer any question that they do not feel comfortable answering, or to choose to end their participation in the study at any time. We do not anticipate any psychological risk that may result from study participants. All measures will be taken to minimize the risk related to the contracting and spreading COVID-19 among any of the researchers or study participants, following the guidelines of the Ministry of Health and the University.

### **Safety and Adverse Events**

All referral processes will be handled by HIAS as follows.

### **CASE MANAGEMENT PROTOCOL AND REFERRAL ROUTES**

At HIAS, we have developed clear pathways and procedures to prevent, identify, and promptly address the needs of all Persons of Concern (PDI), that is, all participants who are directly or indirectly involved with each of our programs. For HIAS Colombia, it is essential to meet the needs of our beneficiaries, especially those who will be part of the Owning Rights and Protection: GBV Prevention, Mitigation, and Response in Colombia project.

This protocol was created to specify the pathways for care and management of cases and needs that may arise during the implementation of the research and that, in turn, represent a risk to the psychosocial well-being and safety of our participants and their families. For example, cases of PDI who are not selected to participate in the EGV, participants who have been randomly assigned to the control group, and/or participants who receive EGV training and express some type of need for care.

#### STEPS FOR CASE MANAGEMENT AND REFERRAL ROUTES

The following describes the procedure designed in conjunction with all strategic areas of HIAS, with the aim of providing clarity on the comprehensive case management and referral pathways we regularly implement as an organization to ensure the protection of our beneficiaries and provide an immediate response to their needs.

HIAS has a robust network of services for the population, as well as referral and counter-referral pathways with other humanitarian organizations and institutional entities to ensure the protection of participants.



Chart 1. Procedure for case management and referrals within the SRI-PRM research project

### Stage 1. Preparation for a situation or need

The HIAS Colombia team prepares to address the needs of IDPs through actions that promote the appropriate approach and management of cases based on a rights-based, gender-based, and age-based approach, which complies with humanitarian principles and prevents actions that cause harm.

In summary, the following strategies will be implemented:

- HIAS staff will be trained to comply with strict confidentiality standards for case management.
- Clear referral pathways to HIAS services are available, and, if required, external referral pathways will be activated with partner organizations and entities.
- HIAS services are implemented in a coordinated and complementary manner. Constant communication channels will be established between the Economic Inclusion area and other HIAS areas to avoid duplication of care, prevent re-victimization of participants, and facilitate access to services.

Additionally, at HIAS, we work closely with government institutions, partner organizations in the territories, the private sector, and refugee communities, promoting local integration and access to rights and services.

### Stage 2. Identification of situations or needs

When needs or situations arise that affect the psychosocial well-being of our IDPs and/or threaten their continued participation in the program, the HIAS Colombia team will be able to respond to the case by activating the corresponding route, depending on whether it is a GBV or MHPSS case.

Likewise, the following strategies will be developed:

- IE Officers and Research Assistants who will be present at the training and data collection spaces will be trained to address any type of situation or need by providing crisis support and Psychological First Aid to individuals experiencing emotional distress, family conflicts, domestic violence, and suicidal thoughts.
- IE Officers will then inform the IDPs about the services available at HIAS (GBV Case Management, Individual Psychosocial Care, and Legal Protection) and will ask each individual if they would like to be referred to any of these services.

## Stage 3. Recording the Situation or Need

When participants express a need to be assisted by HIAS professionals, the needs and/or situation assessment process is activated.

Likewise, the following actions will be carried out:

- Internal referral forms will be used to describe the identified situation, the level
  of risk identified, the priority range under which the case should be addressed,
  and whether the participant's consent is obtained.
- Once the PDI's consent is obtained, the IE Officer will carry out the referral process to the GBV Case Manager or the MHPSS Officer, using the internal case referral forms provided by the MHPSS and GBV department.
- The MHPSS and GBV services at HIAS Colombia conduct risk and needs assessments to determine the support participants require, as well as to negotiate access to additional services with partner organizations. Should external referrals arise, the GBV Case Manager or the MHPSS Officer will be responsible for making them and following up on them.
- The Economic Inclusion Officer will follow up on referrals and will be in contact with the MHPSS Officer or GBV Manager in charge of providing care to the beneficiary.

HIAS Colombia has developed a matrix of physical and psychosocial risks associated with the implementation of the gender-responsive entrepreneurship school program, and has also implemented risk mitigation actions for each situation.

Stage 4. Response to the situation that occurred or need encountered

4. Respuesta a la situación ocurrida o necesidad encontrada

- Cualquier situación de riesgo o necesidad será canalizada por el Oficial de Inclusión Económica, quien deberá remitir a los Oficiales SMAPS y Gestor de casos VBG segun se requiera.
- •Los asistentes de investigación deberán comunicar de manera inmediata al Oficial de Inclusión Económica sobre la situación y este deberá activar la ruta interna de remisión correspondiente.

Once a need for care arises for an IDP, HIAS is able to receive, assist, and manage the case expeditiously and with a survivor-centered approach.

- The Economic Inclusion Specialist will provide technical support and supervision in case management.
- The Economic Inclusion Coordinator will support the team's supervision and ensure proper compliance with the processes. They will also be in close communication with the MHPSS and GBV Coordinators to provide appropriate support for IDPs attending the gender-focused entrepreneurship school.
- It is worth mentioning that HIAS has protocols and/or case analysis committees in which the participant's continued participation is assessed specifically when incidents of risk of gender-based violence occur during the program's implementation.

#### **REFERRAL PROCESS TO INTERNAL HIAS AREAS**

#### REFERRALS TO MHPSS SERVICES

Individual psychosocial care is part of the third-level technical interventions, which are used to stabilize and provide people of interest with ongoing emotional support that promotes daily functioning, stress management, and healthy grieving, and facilitates the identification of flexible coping strategies.

#### **Criteria for Making MHPSS Referrals**

IE Officers will be able to identify each of the criteria necessary to make a referral to the mental health and individual psychosocial care service. In this sense, once the criteria are identified, the internal referral pathway is activated, where the MHPSS Officer receives, assesses, and provides psychosocial care. To make referrals to the MHPSS area, the following criteria must be met:

- Ø The teaching and research staff's willingness to attend a more complex, specialized MHPSS intervention, in this case, Individual Psychosocial Care.
- Ø Frequency: Presence and recurrence of psychosocial indicators (psychological distress)

- Ø Severity: Intensity of psychosocial indicators (severe, moderate, and mild)
- Ø Stage of the survivor's lifespan
- Ø Interference with areas of functioning (personal, family, social, work)
- Ø Low level of adherence to or appropriation of coping mechanisms

The above criteria are evaluated by the SMAPS Officer based on the description of the reason for referral, which must be included in the referral form previously sent by the EI Officer.

#### **Reasons for Case Closure**

For effective case closure in individual psychosocial care, the following conditions must be met:

- Ø There is evidence of a reduction in the occurrence of psychosocial indicators (subjective distress)
- Ø The person shows less irritability and/or aggressive behavior
- Ø The person shows less distress when speaking and recounting something related to their painful experience
- Ø The person returns to enjoying activities they had usually avoided
- Ø The person feels more motivated to talk with others
- Ø The person becomes active in daily activities
- Ø The person seeks more help
- Ø The person reports fewer somatic symptoms
- Ø The person reports having more tools to cope with their problems
- Ø The person shows an increase in their emotional well-being of at least 3 points on the Warwick Scale

Once the MHPSS Officer verifies that there has been a notable improvement in the IDP's psychosocial well-being, they are responsible for finalizing the individual intervention and proceeding to close the case.

## **GBV SERVICE REFERRALS**

Among the services offered by the GBV area, GBV Case Management provides comprehensive support to women, girls, adolescents, survivors, or members of the LGBTQI+ community who are experiencing any type of violence or are at risk of being subjected to violence due to their gender or factors associated with it.

GBV case management is carried out in three modalities: cross-border, emergency, and comprehensive. Case management includes a process for profiling individuals, assessing their GBV risk level, designing an action plan based on specific GBV needs, outlining commitments and objectives for case management. It also includes making the respective internal and

external referrals to services that mitigate the identified needs, conducting case follow-up, and ultimately closing the case. If the IE Officer identifies any risk or situation of violence among participants participating in the EGSE, they may initiate a referral route to the GBV Case Manager, who will receive, assess, and provide management for the specific case. The GBV Officer will provide support to the Case Manager and provide technical guidance while providing care. The GBV Officer will follow the global protocols developed by HIAS for the management of gender-based violence cases, as well as guidelines based on international standards.

## **Criteria for Referrals to GBV Case Management**

In accordance with the GBV Case Management Action Plan, and specifically the needs of the GBV person, referrals are made to the services they require, which we offer both internally and externally.

The criteria defined for referrals to this service are:

Ø Risk of rights violations due to gender

Ø Being abused and/or discriminated against (physically, verbally, financially, and psychologically) and/or humiliated because of their gender

Ø Being a member of the LGBTQ+ community and being subjected to violence (physically, verbally, financially, and psychologically) or perceiving themselves at risk of being subjected to violence due to their gender.

#### **Reasons for Closing GBV Cases**

To proceed with the closure of GBV cases from the case management service, the following conditions must be met:

- Ø Loss of contact with the survivor for more than one month
- Ø Withdrawal from the process by the survivor
- Ø Compliance with objectives within the framework of rights and services management
- Ø Compliance with the maximum of 6 follow-up sessions that can be provided.

Compliance with these conditions is validated by the GBV Case Manager, who also provides the support and follow-up required by the PDI. The GBV Officer provides supervision and technical support for the appropriate handling of all GBV cases.

## **Data analysis**

Quantitative data analysis

Preliminary and descriptive analyses will include: one-way frequency distributions of each survey item and item composite scores, including measures of central tendency (e.g. mean) and variability (e.g. standard deviation) for continuous, approximately normally distributed composite scores. Cronbach's alpha of 0.6 and above will be used as a threshold cut-off to determine the reliability of the composite scores.

We will also model the variation in participants' responses across time. We will test and compute effect sizes for the following hypotheses:

- Directly following program implementation, women who participate in the intervention will exhibit greater improvement in outcomes, compared with women who do not participate in the intervention.
- Three months following the completion of program implementation, women who participate in the intervention will exhibit greater improvement in outcomes, compared with women who do not participate in the intervention.

We plan to test this hypothesis using random coefficient models. The random coefficient model is similar to conducting a difference in difference analysis, but controls and adjusts for additional covariates such as time, taking into account the fact that the data are repeatedly measured or correlated over time. These models incorporate random intercepts and slopes for each research participant based upon the participant's multiple measurements on outcomes captured over time (pre-test versus post-test) (Longford, 1993).

The inclusion of random intercepts and slopes in these analyses renders them random coefficient models, which are also known as mixed effects models (Verbeke & Molenberghs, 2000), multilevel models (Goldstein, 1995), or hierarchical linear models (HLMs) (Bryk & Raudenbush, 2002). All models will include both time-constant demographic (e.g., gender, prior academic achievement and marital status) and time-varying antecedent covariates (e.g., phasing of program implementation).

#### References

- 1. Bryk, A. S., & Raudenbush, S. W. (1992). Hierarchical linear models: Applications and data analysis methods. Sage Publications, Inc.
- 2. Fitzmaurice, G. M., Laird, N. M., & James, H. (2004). Ware. 2004. Applied longitudinal analysis, 3462-3469
- 3. Goldstein, H. (1995). Hierarchical data modeling in the social sciences. Journal of Educational and Behavioral Statistics, 20(2), 201-204.
  - 4. Kabeer, N. (1999). Resources, agency, achievements: Reflections on the measurement of women's empowerment. Development and change, 30(3), 435-464.
- 5. Longford, N. T. (1993). Logistic regression with random coefficients. ETS Research Report Series, 1993(1), i-50.
- 6. Rodríguez Guerrero, E., Nimeh, Z., & Franco Correa, A. (2021). Women's empowerment in Colombia: A multidimensional approach (No. 2021-028). United Nations University-Maastricht Economic and Social Research Institute on Innovation and Technology (MERIT).
- 7. Seff, I., Leeson, K., & Stark, L. (2021). Measuring self-reliance among refugee and internally displaced households: the development of an index in humanitarian settings. *Conflict and Health*, *15*(1), 1-12.
- 8. Trejos Herrera, A., Alarcón, Y., Bahamón Muñetón, M., Vinnacia Alpi, S., González Gutiérrez, O., Llinás Solano, H. y Quevedo Barrios, D. (2023). Validación escala breve de estrategias resilientes. Interdisciplinaria, 40(2), 479-496.
- 9. Molenberghs, G., & Verbeke, G. (2000). Inference for the random effects. Linear Mixed Models for Longitudinal Data, 77-92.

#### Trabajo de campo

#### **Protection of human subjects**

Are you going to work with human subjects?

- Yes
- □ No
- □ Otro:

### Are you going to work with any of these communities?

- LGBTI communities
- Prisoners
- Victims of the armed conflict
- Clinical patients
- Students
- Black communities
- I will not be working with communities
- Other: GBV survivors and women at riskEn caso de trabajar con otra comunidad, por favor mencione cuál.
- Other: Socioeconomically vulnerable women.

#### Conflict of Interest

We encourage you to declare any conflict of interest you believe may affect the project in question. For more information about conflicts of interest, please visit our page.

No competing interests need be disclosed for any of the researchers involved in the study.

### **Ethical Considerations**

In a maximum of 500 words, outline the ethical considerations that will be taken into account in the implementation of the project, clearly identifying at what points in the project's development ethical dilemmas are anticipated and explaining how you plan to avoid or resolve them in your research. Ethical dilemmas may relate to: data collection, handling, and archiving; conflicts of interest; fabrication, falsification, and plagiarism; research with human subjects; animal research; the project's social responsibility; the project's environmental impact; and issues of authorship and funding, among others. If you do not answer this question, the committee will not consider your project.

According to Resolution number 008430 of 1993 of the Colombian Ministry of Health and Social Protection, this is "research without risk", which includes: "studies that employ retrospective documentary research techniques and methods and those in which no intervention or intentional modification of the biological, physiological, psychological or social variables of the individuals participating in the study is carried out, including: review of medical records, interviews, questionnaires and others in which no sensitive aspects of their behaviour are identified or dealt with".

The study is expected to carry minimal risk of loss of confidentiality associated with participation in group discussions, which will be minimized by data confidentiality measures and by using verbal informed consent procedures. Individuals have the option to not participate, or if they choose to participate, to decline to answer any question that they do not feel comfortable answering, or to choose to end their participation in the study at any time. We do not anticipate any psychological risk that may result from study participants. All measures will be taken to minimize the risk related to the contracting and spreading COVID-19 among any of the researchers or study participants, following the guidelines of the Ministry of Health and the University. All focus group and feedback discussions will be conducted in-person.

Additional detailed information on the consenting process and handling of adverse events and referrals can be found in the protocol above.